CLINICAL TRIAL: NCT06014489
Title: A Single Arm Phase II Trial to Assess Cobicistat Boosted Venetoclax in Combination With Azacitidine (sc) in Adult Patients With Newly Diagnosed Acute Myeloid Leukaemia (AML) Who Are Not Considered Candidates for Intensive Treatment Regimens
Brief Title: A Trial to Assess Cobicistat Boosted Venetoclax in Combination With Azacitidine in Adult Patients With Newly Diagnosed AML
Acronym: HO171
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HO171
Record Dates: First submitted 2023-07-04; First posted 2023-08-28 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax; Cobicistat

STUDY DESIGN:
Intervention Model Description: the study consists of a run-in phase and an extension phase
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm arm extension phase (Experimental): prior to the extention phase, there is a run-in phase with (n= 20 patients of 142 total) with the same study scheme, except that cobicistat is added from cycle 2 onwards to the treatment instead of during cycle 1
  Interventions: Drug: azacitidine; Drug: Venetoclax; Drug: Cobicistat

INTERVENTIONS:
Drug: azacitidine — during run-in and extention phase: from Cycle 1 until relapse
Drug: Venetoclax — during run-in and extention phase: from Cycle 1 until relapse
Drug: Cobicistat — during run-in phase: from cycle 2 until relapse
  during extension phase: from cycle 1 until relapse

SUMMARY:
The treatment of older unfit patients with acute myeloid leukemia (AML) is challenging. The hypomethylating agents (HMA) azacitidine and decitabine have relatively mild side effects and have proven to be feasible for the treatment of older patients and patients with co-morbidities. Currently, venetoclax added to an HMA agent is the new standard of treatment. Since this new standard comes with a substantial societal financial burden, there is a rational to optimize the venetoclax dosing schedule. The CYP3A4 inhibitor cobicistat (COBI) can be used to increase venetoclax exposure, thereby allowing to reduce the dose of venetoclax and thus costs substantially.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a patient must meet all of the following criteria:

* Patients with: a diagnosis of AML and related precursor neoplasms according to ICC-2022 classification (excluding acute promyelocytic leukaemia) (appendix A). Patients may have had previous treatment with erythropoiesis stimulating agents (ESA) for an antecedent phase of MDS. ESAs must be stopped at least two weeks before registration.
* Patients 18 years and older who are considered not fit for intensive chemotherapy or who decline the option of intensive chemotherapy.
* WHO performance status 0, 1 or 2 (appendix E).
* Adequate renal and hepatic functions unless clearly disease related as indicated by the following laboratory values:

  * Adequate renal function as demonstrated by a creatinine clearance ≥ 30 mL/min; calculated by the Cockcroft Gault formula or measured by 24 hours urine collection.
  * Serum bilirubin ≤ 3 x upper limit of normal (ULN), unless considered AML-related or due to Gilbert's syndrome.
  * Alanine transaminase (ALT) ≤ 3 x ULN, unless considered AML-related.
* Male subjects who are sexually active, must agree, from Study Day 1 until at least 90 days after the last dose of study drug, to practice the protocol specified contraception. Male subjects must agree to refrain from sperm donation from initial study drug administration through at least 90 days after the last dose of study drug.
* Female subjects must be either postmenopausal defined as: Age >55 years with no menses for ≥12 months, without an alternative medical cause. OR willing and able to use adequate contraception during and until 180 days after the last protocol treatment.
* Written informed consent.
* Patient is capable of giving informed consent.
* Patient agrees not to participate in another interventional study while on treatment without approval of the (co-) Principal Investigator.

Exclusion Criteria:

A patient who meets any of the following criteria cannot be included in this study:

* Acute promyelocytic leukemia.
* Myelodysplastic syndrome (MDS).
* Patients previously treated for AML or MDS (any anti-leukemic therapy including investigational agents; excluding: 1) erythropoiesis stimulating agents (ESAs); 2) hydroxyurea (hydroxyurea is allowed for the control of peripheral leukemic blasts in patients with leukocytosis).
* Diagnosis of any previous or concomitant malignancy is an exclusion criterion:

  * except when the patient successfully completed treatment (chemotherapy and/or surgery and/or radiotherapy) with curative intent for this malignancy at least 24 months prior to registration;
  * except for basal and squamous cell carcinoma of the skin or in situ carcinoma of the cervix.
* Blast crisis of chronic myeloid leukemia.
* Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, pulmonary disease etc.).
* Cardiac dysfunction as defined by:

  * Myocardial infarction within the last 3 months of study entry, or
  * Reduced left ventricular function with an ejection fraction < 40% as measured by MUGA scan or echocardiogram, or
  * Unstable angina or New York Heart Association (NYHA) grade IV congestive heart failure (see Appendix G), or
  * Unstable cardiac arrhythmias.
* History of stroke or intracranial haemorrhage within 6 months prior to registration.
* Symptomatic central nervous system (CNS) leukemia (NO routinely lumbar puncture required to investigate CNS involvement).
* History of non-compliance to medical regimens or considered unreliable with respect to compliance.
* Senile dementia, mental impairment or any other psychiatric disorder that prohibits the patient from understanding and giving informed consent.
* Current concomitant chemotherapy, radiation therapy, or immunotherapy; other than hydroxyurea.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.
* Unreplaceable use of strong inhibitors or inducers of CYP3A or CYP3A/p-GP substrates with a narrow therapeutic window (e.g. cobicistat or ritonavir for HIV treatment). Please check with Appendix I.
* Intolerability, contra-indication or allergy to one of the study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic equivalence of cobicistat boosted venetoclax and unboosted venetoclax (PK cycle 1 vs PK cycle 2).venetoclax and unboosted venetoclax (PK cycle 1 vs PK cycle 2). | 6-8 months
  run-in phase
Overall survival (OS). | 48 months
  extension phase

SECONDARY OUTCOMES:
Venetoclax and cobicistat CL, Cmax, Tmax, Cmin and AUC0-24. | 6-8 months
  run-in phase
Complete remission (CR) rate defined as CR as best response during or at completion of the treatment, as determined by the Investigator, based on the European LeukemiaNet (ELN2022) recommended response criteria (see Appendix B). | 48 months
  extension phase
CR with incomplete hematologic recovery (CRi) rate, based on the European LeukemiaNet (ELN2022) recommended response criteria (see Appendix B). | 48 months
  extension phase
CR and CR with incomplete hematologic recovery (CRi) rate, based on the European LeukemiaNet (ELN2022) recommended response criteria (see Appendix B). | 48 months
  extension phase
CR with partial hematologic recovery (CRh) rate, based on ELN 2022 recommendations. | 48 months
  extension phase
CR and CR with partial hematologic recovery (CRh) rate, based on ELN 2022 recommendations. | 48 months
  extension phase
CR or CR/CRi or CR/CRh without minimal residual disease (flow and or molecular) (CRMRD- or CR/CRiMRD- or CR/CRhMRD-). | 48 months
  extension phase
Morphologic leukemia-free state (MLFS) rate, based on ELN2022 recommendations. | 48 months
  extension phase
Event free survival (EFS). | 48 months
  extension phase
Relapse-free survival (RFS). | 48 months
  extension phase
Incidence and severity of adverse events according to CTCAE version 5.0. | 48 months
  extension phase
Early (30-day and 60-day) mortality (in general, non-leukemic). | 48 months
  extension phase
Time to next cycle, defined as the time from the start of the cycle until the start of the next cycle. | 48 months
  extension phase
OS of AZA/VEN/COBI treated patients in comparison with a real-world data cohort treated during the same time period and monitored by the Dutch Cancer registry. | 48 months
  extension phase
Prognostic/predictive impact of disease-associated genetic changes at diagnosis. | 48 months
  extension phase
Relapse-associated genetic changes (determined at relapse). The average relative dose intensity will be computed and given by categories. The same will be done for treatment deviation. | 48 months
  extension phase
Clonal evolution during treatment. | 48 months
  extension phase
Exposure-response and exposure-toxicity relation of venetoclax in patients with AML. | 48 months
  extension phase
Cost-savings on venetoclax drug costs. | 48 months
  extension phase
Adherence to venetoclax and cobicistat. | 48 months
  extension phase

CONTACTS AND LOCATIONS:
Locations (18):
- Netherlands (18):
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam-OLVG, Amsterdam
  - NL-Amsterdam-VUMC, Amsterdam
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Breda-AMPHIA, Breda
  - NL-Dordrecht-ASZ, Dordrecht
  - NL-Eindhoven-CATHARINA, Eindhoven
  - NL-Eindhoven-MAXIMAMC, Eindhoven
  - NL-Enschede-MST, Enschede
  - NL-Groningen-UMCG, Groningen
  - NL-Leeuwarden-MCL, Leeuwarden
  - NL-Leiden-LUMC, Leiden
  - NL-Maastricht-MUMC, Maastricht
  - NL-Nieuwegein-ANTONIUS, Nieuwegein
  - NL-Nijmegen-CWZ, Nijmegen
  - NL-Rotterdam-ERASMUSMC, Rotterdam
  - NL-Den Haag-HAGA, The Hague
  - NL-Zwolle-ISALA, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — http://www.hovon.nl